CLINICAL TRIAL: NCT06485141
Title: BeSMART Secure Storage Counseling in the Inpatient Setting
Acronym: BeSMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kelsey Gastineau, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 241305
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Firearm Injury; Safety Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Guardians of hospitalized children in the active comparator group will view a brief medication storage safety video produced by Safe Kids.
  Interventions: Behavioral: Safe Kids Medication
- Intervention (Experimental): Guardians of hospitalized children will receive the study intervention, viewing a 3 minute educational video about the importance of secure firearm storage from the Be SMART program. Additionally, a cable gun lock will be offered to families in the intervention group along with a Frequently Asked Questions handout from Be SMART.
  Interventions: Behavioral: Safe Storage Intervention

INTERVENTIONS:
Behavioral: Safe Storage Intervention — Firearm storage information and secure storage device.
  Arms: Intervention
Behavioral: Safe Kids Medication — The Control participants will view a brief medication storage safety video produced by Safe Kids. A Frequently Asked Questions handout on medication safety created by Safe Kids will be available for parents as well.
  Arms: Control

SUMMARY:
Firearm injuries are the leading cause of death for American youth. While most of these deaths are homicides, approximately one third are suicides and 5% are unintentional shootings where a child gains access to an unsecured firearm and unintentionally pulls the trigger injuring or killing themselves or someone else. Secure firearm storage in the home has been shown to significantly reduce the risk of both unintentional shootings and intentional self-harm behavior. Additionally, approximately 75% of the guns that show up on school grounds come from the homes of youth or their family members or friends. Despite evidence that secure storage counseling delivered in the pediatric outpatient setting significantly improves secure storage behavior AND recommendations from the American Academy of Pediatrics to provide secure storage counseling during well child checks, rates of counseling continue to be low. The Be SMART program is aligned with the American Academy of Pediatrics policy statement and recommendations and provides a scalable solution to efficient counseling in the clinical setting. However, except for one single site inpatient study, the efficacy of the Be SMART program has not been formally evaluated in the inpatient pediatric setting.

By rigorously evaluating the efficacy of specific secure storage interventions like Be SMART the investigators can eventually improve counseling frequency with the goal of increasing gun safety behaviors and reducing firearm injuries and deaths in youth.

The investigators hypothesize the Be SMART educational intervention, when delivered in the pediatric inpatient setting, will lead to significant improvement in the primary gun safety behavior endpoint and the secondary endpoint among both gun owners and non-gun owners when compared to control group.

DETAILED DESCRIPTION:
This is a randomized controlled trial, that will utilize computer generated randomization, 1:1 intervention to control group ratio, randomized at the individual patient level. Randomization will occur after informed consent is obtained, before initial survey is administered. The Research Assistant will use computer generated randomization.

There will be 150 subjects per study arm (300 total). The two enrollment sites will each enroll 150 subjects (75 control and 75 intervention) with at least 33% being gun owners. For every 30 subjects enrolled, the site Principal Investigator and Research Assistant will ensure that 10 are gun owners. Once 20 non-owners are enrolled, non-gun owner enrollment will be paused until 10 gun owners are enrolled. This will ensure distribution of gun-owner enrollment over the entire study recruitment period. Enrollment will be ongoing until sample size is reached. Control group will receive an education intervention (video and handout) about the importance of securely storing medications in the home to prevent unintentional ingestions and suicide attempts. This is a multisite trial conducted at Monroe Carell Jr. Children's Hospital and Children's Hospital of Colorado.

During the initial study visit, after screening, enrollment including informed consent, randomization and baseline survey, the participant will either receive the Be SMART intervention (video shown on tablet) with Be SMART postcard sized handout OR the control intervention (SAFE KIDS medication storage video shown on tablet). Immediate post-intervention survey will be completed electronically, and the study visit will conclude.

The study intervention is the viewing of a brief educational video about the importance of secure firearm storage from the Be SMART program. Additionally, a secure storage device (cable gun lock) will be offered to families in the intervention group. A clinician will be available to answer any follow-up questions that study participants may have regarding secure firearm storage.

The control participants will view a brief medication storage safety video produced by SAFE KIDS. A clinician will be available to answer any follow-up questions that study participants may have regarding secure firearm storage. This control video was selected because like secure firearm storage it addresses youth injury risk mitigation and self-harm behavior prevention in the home.

There are two follow-up visits (electronic/phone, no in-person follow-up required): 1-month post-enrollment/intervention delivery and 3 months post-enrollment/intervention delivery. Participants will be contacted via their provided e-mail with a link to the follow-up survey. There will be 3 attempts to contact participants by email. If no response, participants will be contacted by phone, with 3 attempts. If the participants are unable to be reached at this point, they will be considered lost to follow-up.

ELIGIBILITY:
Inclusion Criteria (must meet ALL):

1. Provision of signed and dated informed consent form
2. Caregiver of child hospitalized on a pediatric hospital medicine service aged 0-17
3. English or Spanish speaking caregiver
4. Access to necessary resources for participating in a technology-based intervention follow-up assessments (e-mail and telephone)

Exclusion Criteria:

1. Caregivers of children admitted for firearm injury
2. Caregivers of children with a firearm injury within the last 3 months
3. Caregivers of children admitted with a primary psychiatric diagnosis including suicidal ideation, self-harm, homicidal ideation, aggression, or intentional ingestion
4. Caregivers of children who are admitted to a surgical co-management team

Non-gun owners will be excluded intermittently throughout the enrollment period based on proportion of gun owners enrolled. For every 30 study participants enrolled, 10 must be gun owners. Non-gun owner enrollment will be paused until 10 gun owners are enrolled and this cycle will repeat for every 30 participants enrolled at each study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Secure firearm storage among gun owners | 1 month
  Self-reported secure storage behavior will be the primary endpoint for gun-owners in the sample. Participants will respond to the survey question of "Please share how the majority (meaning more than half) of the guns (such as pistols, revolvers, shotguns, and rifles) in your home/vehicles are stored." with an ordinal scale of storage (Locked and Unloaded, Locked and Loaded, Unlocked and Unloaded, and Unlocked and Loaded) in decreasing order of safety. Responses will be analyzed comparing Locked and Unloaded to the other three choices for a dichotomous measure.
Asking about firearm storage among all participants | 1 month
  Self- report based on the survey question "How often do you ask about the presence of firearms in homes where your child(ren) visits?". Response to the survey question is a Likert scale asking frequency (Never-Rarely - Sometimes - Always - Often).

SECONDARY OUTCOMES:
Asking about firearm storage among all participants | 3 months
  Self- report based on the survey question "How often do you ask about the presence of firearms in homes where your child(ren) visits?". Response to the survey question is a Likert scale of asking frequency (Never-Rarely - Sometimes - Always - Often).

OTHER OUTCOMES:
Firearm Storage Knowledge | 1 month and 3 months
  Caregivers' knowledge and beliefs about firearm storage in the home will be assessed by asking survey questions "It is important for doctors who take care of children to talk to parents/ guardians about safe gun storage.", "It is important for people who have guns to store their firearms with a storage device such as a gun safe or trigger lock" and It is important for parents/guardians to ask if there are any guns in the home, when their child/children go to play in another person's home." with a 5-point Likert scale from Strongly Disagree to Strongly Agree.
Secure firearm storage among gun owners | 3 months
  Self-reported secure storage behavior will be the primary endpoint for gun-owners in the sample. Participants will respond to the survey question of "Please share how the majority (meaning more than half) of the guns (such as pistols, revolvers, shotguns, and rifles) in your home/vehicles are stored." with an ordinal scale of storage (Locked and Unloaded, Locked and Loaded, Unlocked and Unloaded, and Unlocked and Loaded) in decreasing order of safety. Responses will be analyzed comparing Locked and Unloaded to the other three choices for a dichotomous measure.
Locking behavior | 1 month and 3 months
  Self- report at two time points based on the survey question, "Please share how the majority (meaning more than half) of the guns (such as pistols, revolvers, shotguns, and rifles) in your home/vehicles are stored." with an ordinal scale of storage (Locked and Unloaded, Locked and Loaded, Unlocked and Unloaded, and Unlocked and Loaded) in decreasing order of safety. Responses will be analyzed comparing guardians who answered "Locked and Unloaded" or "Locked and Loaded" at follow up to the other two choices for a dichotomous measure.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Gastineau, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No